MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

Date posted to web: 12/05/17

INSTITUTE: National Cancer Institute

STUDY NUMBER: 15-C-0075 PRINCIPAL INVESTIGATOR: Hoyoung Maeng, M.D.

STUDY TITLE: A Randomized, Placebo-Controlled Phase II Study of Multi-Epitope TARP Peptide

Autologous Dendritic Cell Vaccination in Men with Stage D0 Prostate Cancer

Continuing Review Approved by the IRB on 10/16/17 Amendment Approved by the IRB on 12/04/17 (D)

Addendum 1 to 15-C-0075

This addendum provides new information about the study "A Randomized, Placebo-Controlled Phase II Study of Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Men with Stage D0 Prostate Cancer" on which you are enrolled. The information in the consent you signed previously is unchanged.

The NIH Clinical Center Pharmaceutical Development Service (PDS) helps to make the ME TARP DC vaccine used in this study. The PDS was recently closed down by NIH leadership after a vial of contaminated material was discovered on another study just before it was supposed to be given to a research participant. The PDS is undergoing a full review and changes are being made to make sure that processes are in place to prevent anything like this from happening again. The FDA and NIH decided that it might be better and safer to make an exception to the PDS shutdown for some research studies as long as those decisions are made on a case by case or protocol by protocol basis. The ME TARP DC vaccine received one of those exceptions because the parts of the vaccine made by the PDS are just used in the preparation of the vaccine and are never actually given to you, the research participant. Additionally, all of the materials used in making the ME TARP DC vaccine have to pass many tests or they can't be used. Before giving the exception, the FDA and NIH determined that the risk to you from receiving a vaccine that includes the portions made by the PDS, before all of the reviews and changes to the PDS are finished, is extremely low.

• Adult Patient or NIH-2514-1 (07-09)

• Parent, for Minor Patient

P.A.: 09-25-0099

File in Section 4: Protocol Consent (2)

MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 15-C-0075 CONTINUATION: page 2 of 2 pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study | | I have read the explanation about this study | |
| and have been given the opportunity to discuss | | and have been given the opportunity to discuss | |
| it and to ask questions. I hereby consent to | | it and to ask questions. I hereby give | |
| take part in this study. | | permission for my child to take part in this | |
| - | | study. | |
| | | (Attach NIH 2514-2, Minor's Asse | ent, if |
| | | applicable.) | |
| Signature of Adult Patient/ | Date | Signature of Parent(s)/ Guardian | Date |
| Legal Representative | Date | Signature of Farent(s)/ Guardian | Date |
| Legar Representative | | | |
| Print Name | | Print Name | |
| C Child's Voybal Assent (If An | nliaahla) | | |
| C. Child's Verbal Assent (If Applicable) The information in the above consent was described to my child and my child agrees to | | | |
| participate in the study. | | | |
| participate in the study. | | | |
| Signature of Parent(s)/Guardian Date | | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE | | | |
| FROM OCTOBER 16, 2017 THROUGH OCTOBER 15, 2018. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| | | 5 | |
| | | D: (N | |
| Print Name | | Print Name | |

PATIENT IDENTIFICATION

## **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)**

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent